CLINICAL TRIAL: NCT06523920
Title: Protecting Autologous Free Flaps From Ischemia/Reperfusion Damage With Cold Storage: a Randomized Controlled Trial
Brief Title: Protecting Autologous Free Flaps From Ischemia/Reperfusion Damage With Cold Storage.
Acronym: PAFFIRD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cagliari (Other)
Responsible Party: Principal Investigator, Filippo Boriani, Associate Professor, University of Cagliari
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MUR: P2022EEZ8R
Record Dates: First submitted 2024-06-29; First posted 2024-07-26 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Ischemia Reperfusion Injury
Keywords: free flap; microsurgery; cold ischemia
MeSH Terms: conditions — Reperfusion Injury | interventions — Cryopreservation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- UWsolution (Experimental): Flap preserved in UW solution and cold storage during the ischemia time
  Interventions: Device: University of Wisconsin solution + cold storage
- No perfusion (Sham Comparator): Flap without perfusion and cold storage
  Interventions: Other: Unperfused free flap under warm ischemia

INTERVENTIONS:
Device: University of Wisconsin solution + cold storage — Preservation of the free flap with UW solution and cold storage during ischemia time
  Arms: UWsolution
Other: Unperfused free flap under warm ischemia — Traditional processing of the free flap: no perfusion of the flap and warm ischemia (room temperature conservation during ischemia time
  Arms: No perfusion

SUMMARY:
Reconstructive microsurgery allows autologous transplantation of flaps. The procedure causes temporary ischemia. The absence of perfusion and the post-anastomosis reperfusion causes ischemia/reperfusion (I/R) damage and an increased percentage of flap complications associated with the longer duration of the ischemia time. In reconstructive surgery the utilization of preservation solution is very limited. The research hypothesis is that cold storage of free flaps might offer benefits. The present study is a RCT to evaluate the feasibility and safety of a cold preservation (using the UW solution) of the free flaps from I/R damage in oncological microsurgical reconstructions. Blood perfusion will be intraoperatively evaluated through indocyanine green and SPY-DHI.

Moreover, patients' outcomes will be evaluated postoperatively through clinical and radiological examinations, particularly focusing on somatosensory recovery and dental rehabilitation after mandibular reconstruction.

DETAILED DESCRIPTION:
Status of the art Reconstructive microsurgery, via microvascular anastomosis of 0.5 mm to 3 mm vessel diameter, needing an operating microscope, allows autologous transplantation of tissue blocks (flaps) from a donor site to a distant recipient site. The procedure involves temporary ischemia. The absence of perfusion and the post-anastomosis reperfusion causes ischemia/reperfusion (I/R) damage. There is clinical evidence supporting an increased percentage of flap complications associated with the longer duration of the ischemia time. At present, although there are several preservation solutions, for solid organ preservation the University of Wisconsin (UW) solution is still considered the gold standard. Cold storage is also used in autologous liver bench surgery, but not for microvascular reconstruction. Unfortunately, this application of ischemia preservation did not occur in microvascular reconstruction because flaps were considered less prone to damage, having a less functional role, pertaining simply to "filling" or "reshaping". However, this is not the whole truth, if we consider for example the fibula flap, containing an abundance of muscle, which is a vulnerable tissue, and above all the fibula free flap requires a great deal of bone healing, which is necessary for the following dental implants. Moreover, the quality preservation of the original tissues is of paramount clinical relevance if we think about the importance of a soft breast, of a pliable facial reconstruction and, above all, of a functional recovery in a replanted finger, where fibrotic degeneration may cause a functional disaster in terms of range of motion and sensation recovery. To our knowledge, in reconstructive surgery, except for reconstructive transplantation (Vascularized Composite Allotransplantations, VCA), the utilization of preservation solution is very limited.

However, in reconstructive microsurgery and hand/finger replantation, the warm ischemia time can be significantly longer due to flap preparation and difficult implanting within the recipient site, or due to intraoperative technical problems, and some flaps include tissues more vulnerable to warm ischemia time; consequently, it could be useful to use the same procedures employed in VCA to limit I/R injury. A comparative evaluation of the effects of cold preservation of auto-transplanted tissues versus the traditional treatment in which no preservation is performed is non-existing in the medical literature. This lack of scientific knowledge warrants the organization of studies investigating these unexplored aspects of microvascular reconstructive surgical science.

Aims The research hypothesis determining the objectives of this project is that cold static storage of autologous free flaps might offer benefits in terms of flap survival and better preservation of all tissues within the flaps, reducing the incidence of complications, flap shrinkage and the amount of fibrosis induced by I/R damage. Indeed, despite a flow-through and patent microvascular anastomoses, microcirculation and perfusion of the flap can be impaired due to endothelial damage, possibly induced by the I/R traumatic experience that can lead to irreversible fibrosis ending in partial necrosis of the flap and could also explain the significant complication rate (36.1% in head and neck surgery and 35% in breast surgery according to recent studies) in terms of partial flap loss or other early and late complications (Clavien-Dindo grade III), which are more frequent than total flap loss, reported around 2-3% of free tissue transfers in the breast and head and neck regions (2% in breast microsurgical reconstruction and 1-3% in head and neck reconstructions based on published reports). The University of Wisconsin (UW) solution is still considered the gold standard among the preservation solutions in solid organ transplantation as well as in VCA. The UW solution was developed by the surgeon Folkert Belzer and the basic scientist James Southard at the University of Wisconsin in the 1980s and was introduced for clinical use in the United States in 1987. UW solution is characterized by a buffer system (phosphate buffer), with high potassium and low sodium as electrolytes, which mimics the intracellular milieu; in addition, it contains raffinose and lactobionic acid, as osmotic membrane-impermeable agents, molecules that have a large molecular weight (594 and 358 Da) and counteract the transmembranous water shift to prevent cellular edema.

Hydroxyethyl starch was also added as an oncotic substance to prevent expansion of the extracellular space. However, hydroxyethyl starch confers the relatively high viscosity (5.70 cp) to UW solution, which is approximately four times higher than water. Overall the electrolyte composition and the membrane-impermeable macromolecules in UW solution maintain the ionic and osmotic balance during hypothermia. Allopurinol was added as an inhibitor of xanthine oxidase, which blocks the generation of reactive oxygen species (ROS) via the hypoxanthinexanthine- uric acid pathway. The antioxidant glutathione was added to neutralize ROS that are generated during reoxygenation at the time of reperfusion. UW solution also includes adenosine, which serves as a substrate for the resynthesis of ATP on reperfusion. UW solution also omitted Ca2+ because of the extremely low physiological intracellular Ca2+ concentration and the known negative effects of elevated intracellular Ca2+ concentration for cell survival. At present, in literature cold storage for autologous microvascular free tissue transfers has not been reported. Therefore, this project aims to reduce the risks of total and partial free flap failure or fibrotic degeneration and consequent early and late complications, using perfusion of the flaps and their cold storage in UW solution to reduce the I/R damage. Indeed, although the total ischemia time is significantly shorter in autologous free flaps compared to those reported in solid organ transplantation, the longer warm ischemia times sometimes reported in reconstructive surgery should be avoided or somehow neutralized. Moreover, in hand and finger replantation, where surgery is not elective but emergency-based, ischemia times may often be significantly longer.

Sudden circulation interruption alters cellular oxygen and nutrient supply, inducing mitochondrial damage and affecting the metabolic function of the tissues. Reperfusion suddenly restores oxygen and nutrient supply and, following the ischemic time, represents a challenge for the flap tissues that may become particularly sensitive to ROS production. ROS trigger free radical attack to cellular membrane polyunsaturated fatty acids (PUFA) and induce lipid peroxidation, with the formation of unstable fatty acid hydro(pero)xides, eicosanoids, and non-enzymatic (free radical-induced) isoprostanes capable of further propagating free radical reactions thereby extending the damage. I/R damage has a described role in hampering flap integration within the recipient site, its normal and smooth healing with the highst possible degree of similarity to the native preoperative donor tissue. I/R damage determines fibrotic reactions and consequent damage to the neurosensory function due to interference of the scar tissue with the nerve network. In case of mandibular reconstruction, I/R damage is supposed to worsen the quality of bone stock in the reconstructied neomandibula, thereby reducing the possibility of osteointegrated dental implants. Purpose of the study is to evaluate the effect of cold preservation on reconstructive flaps for the breast and head & neck areas, in terms of multiple clinical and radiological endpoints, with a focus on intraoperative evaluation of perfusion, and postoperative neurosensory recovery and quality of the bone in fibula-based mandibular reconstruction, in view of dental implant osteo-integration.

Project The present study is a RCT to evaluate the efficacy of cold preservation of free flaps from I/R damage in post-oncological microsurgical reconstructions. The study design will conform to the CONSORT guidelines for RCTs. The project has been approved by the local IRB. An anonymous database (only patient initials) will be created to record all the included patients' data and it will not be available to the blinded outcomes assessors. The recorded data will be ischemia time (the time between vessel division and reperfusion at the end of microvascular anastomoses), weight of the flap and duration of surgery, patients' demographics, BMI, smoking and comorbidities. Two randomization lists (breast and head & neck) will be created through a randomization list generator, available online (random.org), with a 5 block assignment to Group A (flap preserved in UW solution and cold storage during the ischemia time) and Group B (flap without perfusion and cold storage). The randomization will be kept blinded to the outcome assessors and the radiologists. Once harvested and detached from their donor sites, the flaps of Group A will be flushed with 200 ml UW solution at 4°C into the flap artery within 2 minutes after vessel division.

Following the intra-flap injection of the first 150 ml, the last 50 ml of solution will be used to externally irrigate the outer flap, which will be stored at 4°C during the bench surgery and the anastomoses. Before its reperfusion, the flap will be flushed again through its artery with 0.9% saline solution. The flaps of Group B will be stored at room temperature during the bench surgery and the anastomosis time.

ELIGIBILITY:
Inclusion Criteria:

* Post-oncological mandible reconstruction through fibula free flap,
* Post-oncological soft tissue reconstruction through ALT (Anterior Lateral Thigh) free flap in head and neck region
* Post-oncological breast reconstruction through DIEP (Deep Inferior Epigastric Perforator) and PAP (Profunda femoris Artery Perforator) free flaps.

Exclusion Criteria:

* Malnutrition
* Malabsorption
* Vasculitis
* Pathologies of the connective tissue

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Rate of total flap loss | 1 month
  Frequency of flaps that suffer from complete loss and are removed evaluated through fluorescence after the injection of indocyanine green by means of SPY PHI (Portable Handheld Imager) by Stryker (Kalamazoo, USA),
Rate of partial flap loss | 1 month
  Frequency of flaps that suffer from partial loss and are debrided

CONTACTS AND LOCATIONS:
Overall Officials: Adriana Cordova, Prof, Principal Investigator — University of Palermo

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared with other researchers, they will be kept confidential as per legal requirements

REFERENCES:
- [Background] Dubay D, Gallinger S, Hawryluck L, Swallow C, McCluskey S, McGilvray I. In situ hypothermic liver preservation during radical liver resection with major vascular reconstruction. Br J Surg. 2009 Dec;96(12):1429-36. doi: 10.1002/bjs.6740. PMID 19918862
- [Background] Saeb-Parsy K, Martin JL, Summers DM, Watson CJE, Krieg T, Murphy MP. Mitochondria as Therapeutic Targets in Transplantation. Trends Mol Med. 2021 Feb;27(2):185-198. doi: 10.1016/j.molmed.2020.08.001. Epub 2020 Sep 17. PMID 32952044
- [Background] Hegge JO, Southard JH, Haworth RA. Preservation of metabolic reserves and function after storage of myocytes in hypothermic UW solution. Am J Physiol Cell Physiol. 2001 Sep;281(3):C758-72. doi: 10.1152/ajpcell.2001.281.3.C758. PMID 11502553
- [Background] Coriddi M, Myers P, Mehrara B, Nelson J, Cordeiro PG, Disa J, Matros E, Dayan J, Allen R, McCarthy C. Management of postoperative microvascular compromise and ischemia reperfusion injury in breast reconstruction using autologous tissue transfer: Retrospective review of 2103 flaps. Microsurgery. 2022 Feb;42(2):109-116. doi: 10.1002/micr.30845. Epub 2021 Dec 2. PMID 34854501
- [Background] Suh JD, Sercarz JA, Abemayor E, Calcaterra TC, Rawnsley JD, Alam D, Blackwell KE. Analysis of outcome and complications in 400 cases of microvascular head and neck reconstruction. Arch Otolaryngol Head Neck Surg. 2004 Aug;130(8):962-6. doi: 10.1001/archotol.130.8.962. PMID 15313867
- [Background] Peeters WJ, Nanhekhan L, Van Ongeval C, Fabre G, Vandevoort M. Fat necrosis in deep inferior epigastric perforator flaps: an ultrasound-based review of 202 cases. Plast Reconstr Surg. 2009 Dec;124(6):1754-1758. doi: 10.1097/PRS.0b013e3181bf7e03. PMID 19952630
- [Background] Heidekrueger PI, Moellhoff N, Horch RE, Lohmeyer JA, Marx M, Heitmann C, Fansa H, Geenen M, Gabka CJ, Handstein S, Prantl L, von Fritschen U. Overall Complication Rates of DIEP Flap Breast Reconstructions in Germany-A Multi-Center Analysis Based on the DGPRAC Prospective National Online Registry for Microsurgical Breast Reconstructions. J Clin Med. 2021 Mar 2;10(5):1016. doi: 10.3390/jcm10051016. PMID 33801419
- [Background] Nagel TH, Hayden RE. Mayo Clinic Experience with Unfavorable Results After Free Tissue Transfer to Head and Neck. Clin Plast Surg. 2016 Oct;43(4):669-82. doi: 10.1016/j.cps.2016.05.005. Epub 2016 Jun 22. PMID 27601391
- [Background] Belzer FO, Southard JH. Principles of solid-organ preservation by cold storage. Transplantation. 1988 Apr;45(4):673-6. doi: 10.1097/00007890-198804000-00001. No abstract available. PMID 3282347
- [Background] Morrow JD, Roberts LJ. The isoprostanes: unique bioactive products of lipid peroxidation. Prog Lipid Res. 1997 Mar;36(1):1-21. doi: 10.1016/s0163-7827(97)00001-5. PMID 9373618
- [Background] Banni S, Montisci R, Sanfilippo R, Finco G, Sanna D, Giordano E, Murru E, Cordeddu L, Carta G, Banni D, Marchi A. Physiological response to lipid peroxidation in ischemia and reperfusion during carotid endarterectomy. Lipids Health Dis. 2010 Apr 21;9:41. doi: 10.1186/1476-511X-9-41. PMID 20409338
- [Background] Iannone A, Petroni A, Murru E, Cordeddu L, Carta G, Melis MP, Bergamini S, Casa LD, Cappiello L, Carissimi R, O'Shea M, Bell D, De Santis E, Banni S. Impairment of 8-iso-PGF(2ALPHA) isoprostane metabolism by dietary conjugated linoleic acid (CLA). Prostaglandins Leukot Essent Fatty Acids. 2009 May-Jun;80(5-6):279-87. doi: 10.1016/j.plefa.2009.02.008. Epub 2009 Apr 28. PMID 19403295
- [Background] Ebner JJ, Mehra T, Gander T, Schumann P, Essig H, Zweifel D, Rucker M, Slankamenac K, Lanzer M. Novel application of the Clavien-Dindo classification system and the comprehensive complications index(R) in microvascular free tissue transfer to the head and neck. Oral Oncol. 2019 Jul;94:21-25. doi: 10.1016/j.oraloncology.2019.05.005. Epub 2019 May 9. No abstract available. PMID 31178208
- [Background] Katsuragi Y, Kayano S, Akazawa S, Nagamatsu S, Koizumi T, Matsui T, Onitsuka T, Yurikusa T, Huang WC, Nakagawa M. Mandible reconstruction using the calcium-sulphate three-dimensional model and rubber stick: a new method, 'mould technique', for more accurate, efficient and simplified fabrication. J Plast Reconstr Aesthet Surg. 2011 May;64(5):614-22. doi: 10.1016/j.bjps.2010.08.010. Epub 2010 Sep 29. PMID 20884306
- [Background] Zhang L, Liu Z, Li B, Yu H, Shen SG, Wang X. Evaluation of computer-assisted mandibular reconstruction with vascularized fibular flap compared to conventional surgery. Oral Surg Oral Med Oral Pathol Oral Radiol. 2016 Feb;121(2):139-48. doi: 10.1016/j.oooo.2015.10.005. Epub 2015 Oct 23. PMID 26792754
- [Background] Bjordal K, de Graeff A, Fayers PM, Hammerlid E, van Pottelsberghe C, Curran D, Ahlner-Elmqvist M, Maher EJ, Meyza JW, Bredart A, Soderholm AL, Arraras JJ, Feine JS, Abendstein H, Morton RP, Pignon T, Huguenin P, Bottomly A, Kaasa S. A 12 country field study of the EORTC QLQ-C30 (version 3.0) and the head and neck cancer specific module (EORTC QLQ-H&N35) in head and neck patients. EORTC Quality of Life Group. Eur J Cancer. 2000 Sep;36(14):1796-807. doi: 10.1016/s0959-8049(00)00186-6. PMID 10974628
- [Background] Hassan SJ, Weymuller EA Jr. Assessment of quality of life in head and neck cancer patients. Head Neck. 1993 Nov-Dec;15(6):485-96. doi: 10.1002/hed.2880150603. PMID 8253555
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Background] Draaijers LJ, Tempelman FR, Botman YA, Tuinebreijer WE, Middelkoop E, Kreis RW, van Zuijlen PP. The patient and observer scar assessment scale: a reliable and feasible tool for scar evaluation. Plast Reconstr Surg. 2004 Jun;113(7):1960-5; discussion 1966-7. doi: 10.1097/01.prs.0000122207.28773.56. PMID 15253184
- [Background] Pusic AL, Klassen AF, Scott AM, Klok JA, Cordeiro PG, Cano SJ. Development of a new patient-reported outcome measure for breast surgery: the BREAST-Q. Plast Reconstr Surg. 2009 Aug;124(2):345-353. doi: 10.1097/PRS.0b013e3181aee807. PMID 19644246
- [Background] Jang S, Graffy PM, Ziemlewicz TJ, Lee SJ, Summers RM, Pickhardt PJ. Opportunistic Osteoporosis Screening at Routine Abdominal and Thoracic CT: Normative L1 Trabecular Attenuation Values in More than 20 000 Adults. Radiology. 2019 May;291(2):360-367. doi: 10.1148/radiol.2019181648. Epub 2019 Mar 26. PMID 30912719
- [Background] Tayyab SJ, Adrada BE, Rauch GM, Yang WT. A pictorial review: multimodality imaging of benign and suspicious features of fat necrosis in the breast. Br J Radiol. 2018 Dec;91(1092):20180213. doi: 10.1259/bjr.20180213. Epub 2018 Jul 31. PMID 29987981
- [Result] Lee KT, Lee JE, Nam SJ, Mun GH. Ischaemic time and fat necrosis in breast reconstruction with a free deep inferior epigastric perforator flap. J Plast Reconstr Aesthet Surg. 2013 Feb;66(2):174-81. doi: 10.1016/j.bjps.2012.09.020. Epub 2012 Oct 25. PMID 23102871
- [Result] Marre D, Hontanilla B. Increments in ischaemia time induces microvascular complications in the DIEP flap for breast reconstruction. J Plast Reconstr Aesthet Surg. 2013 Jan;66(1):80-6. doi: 10.1016/j.bjps.2012.08.024. Epub 2012 Sep 13. PMID 22981497
- [Result] Forni E, Meriggi F. Bench surgery and liver autotransplantation. Personal experience and technical considerations. G Chir. 1995 Oct;16(10):407-13. PMID 8588982